CLINICAL TRIAL: NCT00483184
Title: Phase II Study, Evaluation of Low Dose Natural Human Interferon Alpha Administered by the Oral Mucosal Route in the Treatment of Behçet's Disease
Brief Title: Low Dose Interferon Alpha Treatment for Oral Ulcers of Behcet's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nobel Pharmaceuticals (Industry)
Collaborators: Ainos, Inc. (f/k/a Amarillo Biosciences Inc. (Industry)
Responsible Party: Hasan Zeytin, Nobel Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 04HUBD01
Record Dates: First submitted 2007-06-05; First posted 2007-06-06 (Estimated); Results first posted 2009-06-16 (Estimated); Last update posted 2009-06-16 (Estimated); Status verified 2009-04

CONDITIONS: Behcet Syndrome; Behcet Disease; Mucocutaneous Ulceration
MeSH Terms: conditions — Behcet Syndrome | interventions — Interferon-alpha

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Placebo Comparator): (placebo)0 IU IFNa
  Interventions: Biological: Veldona,
- 2 (Experimental): (Veldona)500 IU IFNα bid
  Interventions: Biological: Veldona,
- 3 (Experimental): (Veldona)1000 IU IFNα bid
  Interventions: Biological: Veldona,

INTERVENTIONS:
Biological: Veldona, — Very low dose oral natural human interferon alpha lozenges

SUMMARY:
The purpose of this study is to determine the safety and efficacy of natural human interferon alpha (IFN alpha) on size, number, incidence and pain of oral ulcers associated with Behçet's Disease (BD).

DETAILED DESCRIPTION:
Behçet's disease is a severe chronic relapsing inflammatory disorder marked by oral and genital ulcers, uveitis and skin lesions, as well as varying multisystem involvement including the joints, blood vessels, central nervous system, and gastrointestinal tract. Oral ulcers are the initial symptom for most of Behçet's cases and are the single manifestation of the disease required for an official diagnosis, along with two other hallmark symptoms.

Ninety (90) patients will be enrolled in a randomized, parallel, double-blind, placebo-controlled study to evaluate the effectiveness of low dose natural human IFN α administered by the oral mucosal route in reducing the number, size, incidence and pain of oral ulcers in patients with Behçet's disease.

The clinical trial will consist of 3 groups of patients randomized in a 1:1:1 ratio to twice daily receive 2 lozenges containing 500 IU IFN α(2,000 IU daily, n=30), one active (500 IU) and one placebo lozenge (1,000 IU daily, n=30) or 2 placebo lozenges (n=30). Subjects will be monitored weekly over an initial 4 weeks of treatment and then bi-weekly over an additional 8 weeks of treatment. Medication will be self-administered as 2 lozenges taken twice daily (morning and evening). Oral lesions will be counted and measured at each study visit, and patients will answer a series of questionnaires. Results will be subjected to statistical analysis at the completion of the study, with change in total ulcer burden of a patient, a measurement of the total oral mucosal surface area involved with ulcerous lesions at each visit, serving as the primary endpoint. The total ulcer burden from each treated visit will be compared to the baseline total ulcer burden and the amount of change determined. Patients with a 75% decrease in total ulcer burden will be considered responders.

ELIGIBILITY:
Inclusion Criteria:

* Is a male or a non-pregnant, non-lactating female.
* Has a history and clinical presentation consistent with a diagnosis of Behçet's Disease and meets International Study Group criteria (Appendix B).
* Has a history of oral ulcers for at least 12 months.
* Has a history of monthly episodes of multiple oral ulcers.
* Has the presence of at least 2 oral ulcers at study entry, both of which are accessible to measurement, with a total diameter of at least 4 mm.
* Has signed an IRB approved subject consent form.
* Has completed all screening procedures satisfactorily, is deemed to be an acceptable subject and is otherwise eligible for entry into the study.
* Is willing and able to comply with the protocol.

Exclusion Criteria:

* Has a severe, acute, or chronic systemic disease other than Behçet's Disease such as congestive heart failure, hepatic failure, renal failure, Systemic Lupus Erythematosus (SLE), Stevens-Johnson syndrome, ulcerative colitis, cancer, leukemia, diabetes, AIDS or ARC, or any other condition for which they are immunocompromised.
* Is under active treatment for dental conditions, such that multiple dental office visits would be required during the study period, or presents with oral conditions which are not thought to be related to Behçet's Disease and, in the judgment of a qualified dentist, will require treatment during the study period.
* Is suffering from any medical condition other than Behçet's Disease known to cause oral ulcerations, such as erosive lichen planus, benign mucous membrane pemphigoid, SLE, Crohn's disease, Reiter's syndrome, or AIDS.
* Has an eating disorder and/or psychiatric illness requiring treatment.
* Has hypersensitivity to interferon-alpha.
* Is a pregnant or lactating female, or is of childbearing potential and is not using a medically acceptable contraceptive method throughout the study.
* Has had previous exposure to any parenteral interferon therapy.
* Has had exposure to IFNα lozenges within 30 days of screening.
* Has had exposure to thalidomide within 30 days of screening.
* Has had exposure to methotrexate within 30 days of screening.
* Has had exposure to any immune-suppressive medication within 30 days of screening.
* Has a history of, or is currently exhibiting, any disease or condition which, in the opinion of the Principal Investigator, would place the subject at increased risk during study therapy.
* Has any abnormality in a hematological or biochemical variable which, in the opinion of the Principal Investigator, would place the subject at increased risk during study therapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2006-04; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hasan Yazici, MD, Study Director — Istanbul University Cerrahpaşa Medical School; Cem Mat, MD, Principal Investigator — Istanbul University Cerrahpasa Medical School; Cengiz Korkmaz, MD, Principal Investigator — Osmangazi University Medical School; Ayhan Dinc, MD, Principal Investigator — Gülhane Military Medical School; Ahmet Gul, MD, Principal Investigator — İstanbul University Istanbul Medical School
Locations (4):
- Turkey (Türkiye) (4):
  - Gulhane Military Medical School, Ankara
  - Osmangazi University Medical School, Dept of Rheumatology, Eskişehir
  - Istanbul University Cerrahpasa Medical School Department of Internal Medicine, Istanbul
  - Istanbul University Istanbul Medical School, Istanbul

REFERENCES:
- [Derived] Kilic H, Zeytin HE, Korkmaz C, Mat C, Gul A, Cosan F, Dinc A, Simsek I, Sut N, Yazici H. Low-dose natural human interferon-alpha lozenges in the treatment of Behcet's syndrome. Rheumatology (Oxford). 2009 Nov;48(11):1388-91. doi: 10.1093/rheumatology/kep237. Epub 2009 Aug 28. PMID 19717547

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eighty four Behcet's Disease patients were followed at the rheumatology or dedicated BS outpatient clinics of 4 medical schools in Turkey.
Pre-assignment Details: Consecutive patients aged 18-75 fulfilling Behçet's disease International Study Group criteria (16) with the presence of active oral ulcers (OU) within the previous year were included. A further requirement was the presence of at least 2 OU accessible to measurement and with a total diameter of at least 4 mm.
Groups:
- 1: (placebo)0 IU IFN alpha
Period: Overall Study
Arm/Group | 1 | 2 | 3
Started | 27 | 31 | 26
Completed | 22 | 27 | 23
Not Completed | 5 | 4 | 3
Not completed — Withdrawal by Subject | 2 | 2 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Adverse Event | 1 | 2 | 2
Not completed — Protocol Violation | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 | 2 | 3 | Total
Number analyzed (Participants) | 27 | 31 | 26 | 84
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 27 | 31 | 26 | 84
  >=65 years | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 36 (8.6) | 37 (10.2) | 36 (9.4) | 37 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 19 | 59
  Male | 7 | 11 | 7 | 25
Region of Enrollment [Number; unit: participants]
  Turkey | 27 | 31 | 26 | 84

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Patients Experiencing a Sustained Response for Each Treatment Arm.
Description: A patient with a 75% or greater decrease in total OU for three visits was considered a "sustained responder".
Time Frame: (0-12 weeks)
Measure: Number; unit: patients with sustained response
Arm/Group | 1 | 2 | 3
Number analyzed (Participants) | 22 | 27 | 23
patients with sustained response | 13 | 10 | 12
Statistical Analysis 1: Comparison: 1 vs 2 vs 3; Results were expressed as mean or number. Normal distributed data among the treatment groups were compared by One-way ANOVA test, non-normal distributed data were compared by Kruskal Wallis test, and then Bonferroni post-hoc test was used for multiple comparisons. Differences from baseline within treatment groups were evaluated by repeated measures ANOVA test for normal distributed data, Freidman test for non-normal distributed data; Test type: Superiority or Other; p = 0.404, ANOVA

2. Secondary Outcome: Time to Initial Response, Oral Ulcer Sustained Response, Oral Ulcer Recurrence, Time to Recurrence, Pain Associated With Oral Lesions, General Well-Being, Safety
Time Frame: 12 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | 1 | 2 | 3
Serious Adverse Events (participants affected / at risk) | 0 | 1 | 0
Other Adverse Events (participants affected / at risk) | 2 | 5 | 2
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | 1 | 2 | 3
cervical intraepithelial neoplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/0 (0) | 1/1 (1) | 0/0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk (number of events):
Term (organ system) | 1 | 2 | 3
headache (General disorders) | 2/2 (2) | 4/4 (6) | 2/2 (2)
nausea (Gastrointestinal disorders) | 0/0 (0) | 2/2 (2) | 0/0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less